CLINICAL TRIAL: NCT06021379
Title: Post-marketing Surveillance for Evaluation of AryoTrust Safety in Iranian HER2-positive Breast Cancer Patients Undergoing Adjuvant Chemotherapy Regimens
Brief Title: AryoTrust® (Trastuzumab) Safety Study
Status: Completed | Type: Observational
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRA.ARY.FH.95.IV
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Trastuzumab; Safety; AryoTrust; Breast Cancer; Adjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AryoGen Pharmed Trastuzumab: AryoTrust is given at dosing of 6 mg/m2 after adjuvant chemotherapy completion every 3 weeks for 9 cycles.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — AryoTrust (AryoGen Pharmed Trastuzumab) is given at a dosing of 6 mg/m2 after adjuvant chemotherapy completion every 3 weeks for 9 cycles.
  Other Names: AryoTrust

SUMMARY:
This study was a phase IV, observational, multicenter, single-arm, open-label, post-marketing surveillance study for the assessment of AryoTrust safety in Iranian HER2-positive breast cancer patients undergoing adjuvant chemotherapy regimens.

DETAILED DESCRIPTION:
The present study is an observational, multicenter, non-interventional, single-arm, open-label PMS study conducted in Iran. No control groups are included in the study design.

The objective of this PMS study is to monitor and assess the safety of AryoTrust in patients with non-metastatic HER2-positive breast cancer in adjuvant setting over a period of 27 weeks.

Treatment with AryoTrust in this study is defined as the administration of 6mg/kg AryoTrust, every 3 weeks during the 27 weeks of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER2-positive breast cancer undergoing adjuvant chemotherapy regimens

Exclusion Criteria:

* Patients who had received Trastuzumab as part of their therapy or were not candidates for treatment continuation after adjuvant chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 597 Iranian patients diagnosed with HER2-positive breast cancer who underwent adjuvant chemotherapy regimens with AryoTrust were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety by incidence, severity, seriousness and causality relationship of reported AEs | up to 27 weeks
  Safety assessment, including the incidence of any AEs, laboratory results and assessment of tolerability as evaluated by infusion-related reactions. All AEs were classified based on the Medical Dictionary for Regulatory Activities (MedDRA Desktop Browser 4.0 Beta) terms as System Organ Class (SOC) and Preferred Term (PT). All the reported events were graded according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Moreover, seriousness of AEs was assessed according to International Council for Harmonisation (ICH-E2B) guidelines. The causality relation was assessed based on the World Health Organization (WHO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Fatemeh Homaee Shandiz, Prof., Principal Investigator — Radiooncology Department, school of Medicine, Mashhad University of Medical Sciences
Locations (15):
- Iran (15):
  - 5th Azar Hospital, Gorgan
  - Milad Hospital, Isfahan
  - Mahdieh Clinic, Kermanshah
  - Hashemi Nezhad Hospital, Mashhad
  - Imam Reza Hospital, Mashhad
  - Omid Hospital, Mashhad
  - Sadra Clinic, Qom
  - Vasei Hospital, Sabzawār
  - Namazi Hospital, Shiraz
  - Valiasr Hospital, Tabriz
  - Imam Hussein Hospital, Tehran
  - Mahdiyeh Hospital, Tehran
  - Shahid Fayaz-Bakhsh Hospital, Tehran
  - Shohadaye Tajrish Hospital, Tehran
  - Omid Hospital, Urmia

REFERENCES:
- [Derived] Zahedi F, Jafari A, Nasiri Motlagh B, Hamedi SH, Salek R, Khandoozi S, Farshchian N, Shahidsales S, Mafi AR, Hosseini S, Amouheidari A, Varshoee Tabrizi F, Khanjani N, Ahmadloo N, Dayyani M, Khodabakhshi R, Mojahed MM, Keshvari M, Fazl Ersi M, Mirsadraee M, Izadpanahi P, Saadipoor A, Nasrollahi H, Anbiaee R, Emadi Torghabeh A, Keramati A, Amiran SA, Bayat Mokhtari N, Taghizadeh Kermani A, Anvari K, Sadeghi Ivari M, Dayani M, Amirabadi A, Saeidi Saedi H, Sabzvari A, Kafi H, Homaei Shandiz F. Safety evaluation of the trastuzumab biosimilar in Iranian women with HER2-positive breast cancer undergoing adjuvant chemotherapy: a post-marketing surveillance. Expert Opin Drug Saf. 2024 Aug 1:1-6. doi: 10.1080/14740338.2024.2385483. Online ahead of print. PMID 39076099